CLINICAL TRIAL: NCT07146126
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase IIb/III Study to Assess the Efficacy and Safety of PG-011 Nasal Spray in Adults With Moderate to Severe Seasonal Allergic Rhinitis
Brief Title: A Phase III Study to Assess the Efficacy and Safety of PG-011 Nasal Spray in Adults With Moderate to Severe Seasonal Allergic Rhinitis
Acronym: Pumecitinib
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Prime Gene Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PG-011-SAR-301(phase III)
Record Dates: First submitted 2025-07-25; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-07

CONDITIONS: Seasonal Allergic Rhinitis; SAR
Keywords: SAR; PG-011; Seasonal Allergic Rhinitis; Pumecitinib
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PG-011 nasal spray 0.6%(twice daily) (Experimental): 2 sprays in each nostril, twice daily for 14-day treatment period.
  Interventions: Drug: PG-011 nasal spray 0.6%(twice daily)
- Vehicle nasal spray(twice daily) (Placebo Comparator): 2 sprays in each nostril, twice daily for 14-day treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PG-011 nasal spray 0.6%(twice daily) — 2 sprays in each nostril, twice daily for 14-day treatment period.
  Other Names: Pumecitinib nasal spray
  Arms: PG-011 nasal spray 0.6%(twice daily)
Drug: Placebo — 2 sprays in each nostril, twice daily for 14-day treatment period.
  Other Names: Vehicle of Pumecitinib nasal spray
  Arms: Vehicle nasal spray(twice daily)

SUMMARY:
The study is a multicenter, randomized, double-blind, placebo-controlled seamless and adaptive-designed phase IIb/III study encompassing a phase IIb and a phase III component, phase IIb is a dose-ranging part and has been done, and phase III is a pivotal study part which is registered this time.

The goal of this phase III study is to evaluate the efficacy, safety, and pharmacokinetics of PG-011 nasal spray for treating adults with moderate to severe seasonal allergic rhinitis (SAR). Investigators will compare PG-011 nasal spray to a placebo (a look-alike substance that contains no drug) to see if PG-011 nasal spray works to treat moderate to severe seasonal allergic rhinitis

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled clinical study in adults participants aged from 18 to 65 years old (including threshold) with moderate to severe SAR. Approximately 600 participants will be randomized assigned to one of the 2 following groups in a 2:1 ratio.

PG-011 nasal spray 0.6% (1.2mg Pumecitinib) administered twice daily. PG-011 placebo nasal spray 0% (0 mg Pumecitinib) administered twice daily. Participants will receive blinded study treatment for 14 days followed by 21 days safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 65 (including threshold).
2. Reflective total nasal symptom score ( rTNSS) score≥ 6 and retrospective nasal obstruction ≥ 2 on the day of screening visit, D-4 and D1. Meanwhile, the baseline average rTNSS score(Calculated as the average of rTNSS score of D-3, D-2, D-1 morning, D-1 evening, and D1 morning) ≥ 6
3. History of SAR for at least 2 years. and positive results for any local allergen in the current season tested by either the skin prick test (SPT) (where the wheal diameter is at least 5 mm larger than that of the negative control) or the serum - specific IgE (sIgE) test (the sIgE test results obtained within ≤ 1 year before random enrollment are acceptable).
4. Willingness to avoid pregnancy or fathering children from the signing of the informed consent form until three month after after the end of the study.
5. Willing to sign the informed consent form and abide by the research protocol.

Exclusion Criteria:

1. Participants are diagnosed of active or latent tuberculosis infection.
2. Participants are diagnosed of moderate to severe asthma.
3. Participants who had active pulmonary diseases or infections, upper respiratory tract infections or sinus infections within 2 weeks before screening, and/or those who had respiratory infections during the lead-in period.
4. Participants received nasal or sinus surgery within 3 months before screening or had nasal trauma that had not fully healed.
5. Any nasal mucosal erosion, nasal septal ulcer or nasal septal perforation, as judged by the investigator, may affect the deposition of drugs in the intranasal, such as acute or chronic sinusitis, drug-induced rhinitis, nasal polyps, etc.
6. Participants has ocular herpes simplex or other ocular infections (except seasonal allergic conjunctivitis).
7. Participants with facial or systemic fungal, bacterial, viral or parasitic infections, or oral infections that had not been cured and still required continuous treatment within 4 weeks before screening.
8. Participants have severe diseases such as central nervous system, respiratory system, liver, kidney, gastrointestinal tract, urinary system, endocrine system or blood system, which may affect the judgment of efficacy and safety .
9. Participants who were infected with human immunodeficiency virus (HIV) at the time of screening, those in the active stage of hepatitis C virus (HCV) infection, those in the active stage of hepatitis B virus (HBV) infection (HBV - DNA > 2000 IU/mL or 10⁴ copies/mL), or those with positive Treponema pallidum antibody indicating an active stage of infection.
10. Any drug treatments before lead-in period, such as use of nasal or systemic decongestants and anticholinergic drugs within 3 days, use of antihistamines such as cetirizine, fexofenadine, and loratadine within 5 days, systemic use of glucocorticoids within 4 weeks, mast cell stabilizers, tricyclic antidepressants, and leukotriene receptor antagonists within 2 weeks, and use of anti - allergic Chinese herbal medicines within 2 weeks, use of anti-interleukin-4 receptor α subunit (IL-4Rα) monoclonal antibody such as thymic matrix lymphopoietin (TSLP) monoclonal antibody, anti-IgE monoclonal antibody, other monoclonal antibody, or other biologics within 10 weeks or 5 half-lives (whichever is longer).
11. During the trial, participants who cannot stop using JAK inhibitors, tricyclic antidepressants, glucocorticoids, decongestants, antihistamines (except loratadine, which is a rescue drug required during the treatment), leukotriene receptor antagonists, mast cell stabilizers (including sodium cromoglycate, nedocromil sodium, tetrazolium chromone, nedocromil sodium, pemirolast potassium, and tranilast, etc.), anticholinergic drugs, anti - allergic Chinese herbal medicines, and those who cannot stop using nasal irrigation.
12. Participants who have undergone desensitization therapy or received immunotherapy within 6 months prior to screening.
13. Participants who are known or judged by the investigator to potentially have an allergic reaction to the active ingredients or excipients of the investigational drug.
14. Participants who have a history of intolerance to intranasal administration.
15. Participants who plan to travel outside the local area for 2 consecutive days or more during the trial.
16. Participants who have participated in other clinical studies of investigational drugs or medical devices within 3 months prior to screening and have used investigational products.
17. Participants who have a history of drug abuse or alcoholism within 1 year prior to screening
18. Female participants who are breastfeeding or pregnant at the time of screening
19. Reproductive - age participants (male or female) who plan to become pregnant, breastfeed, or donate sperm/eggs during the study or within 1 month after the study ends
20. Any other condition that, in the opinion of the investigator or sponsor, makes the subject unsuitable for participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in average retrospective Total Nasal Symptom Score (rTNSS) over the 14-day treatment period | Up to Day 14
  The reflective Total Nasal Symptom Score (rTNSS) was assessed by 12-hour reflective scoring (AM, PM) of the severity of four nasal symptoms (rhinorrhea, sneezing, nasal congestion, nasal itching). Scores ranged from 0 (no signs/symptoms evident) to 3 (severe signs/symptoms that is hard to tolerate). The rTNSS was calculated as the sum of the subject-reported severity scores for nasal symptoms, and value ranged from 0 (no signs/symptoms evident) to 12 (severe signs/symptoms that is hard to tolerate). Higher scores indicate more severe nasal symptoms, while lower scores indicate less severe nasal symptoms.

SECONDARY OUTCOMES:
Percent change from baseline in average retrospective Total Nasal Symptom Score (rTNSS) over the 14-day treatment period | Up to Day 14
  The reflective Total Nasal Symptom Score (rTNSS) was assessed by 12-hour reflective scoring (AM, PM) of the severity of four nasal symptoms (rhinorrhea, sneezing, nasal congestion, nasal itching). Scores ranged from 0 (no signs/symptoms evident) to 3 (severe signs/symptoms that is hard to tolerate). The rTNSS was calculated as the sum of the subject-reported severity scores for nasal symptoms, and value ranged from 0 (no signs/symptoms evident) to 12 (severe signs/symptoms that is hard to tolerate). Higher scores indicate more severe nasal symptoms, while lower scores indicate less severe nasal symptoms. Percent change is calculated as (Change from baseline / Baseline result *100).
Change and percent change from baseline in average instantaneous Total Nasal Symptom Score (iTNSS) over the 14-day treatment period | Up to Day 14
  The instantaneous Total Nasal Symptom Score (iTNSS) was assessed by instantaneous symptom severity of four nasal symptoms (rhinorrhea, sneezing, nasal congestion, nasal itching). Scores ranged from 0 (no signs/symptoms evident) to 3 (severe signs/symptoms that is hard to tolerate).The iTNSS was calculated as the sum of the subject-reported severity scores for nasal symptoms, and value ranged from 0 (no signs/symptoms evident) to 12 (severe signs/symptoms that is hard to tolerate). Higher scores indicate more severe nasal symptoms, while lower scores indicate less severe nasal symptoms. Percent change is calculated as (Change from baseline / Baseline result *100).
Change and percentage change from baseline in average retrospective Ocular Symptom Total Score (rTOSS) over the 14-day treatment period | Up to Day 14
  The reflective Ocular Symptom Total Score (rTOSS) was assessed by 12-hour reflective scoring (AM, PM) of the severity of three rocular symptoms (itching/burning, tearing/watering, and redness).Scores ranged from 0 (no signs/symptoms evident) to 3 (severe signs/symptoms that is hard to tolerate). . The Total Ocular Symptom Score (TOSS) ranged from 0 to 9. Higher scores indicate more severe ocular symptoms, while lower scores indicate less severe ocular symptoms. Percent change is calculated as (Change from baseline / Baseline result *100).
Change and percent change from baseline in average instantaneous ocular symptom score (iTOSS) over 14-day treatment period | Baseline and Day 14
  The instantaneous Total ocular Symptom Score is a scale used to measure ocular symptom severity based on how the participant was feeling just before taking each dose of study medication. Scores ranged from 0 to 9, and calculated as the sum of participant's scoring of three individual ocular symptoms (itching/burning, tearing/watering, and redness) on a 0 to 3 categorical severity scale (0=absent, 1=mild, 2=moderate, and 3=severe).
  Percent change is calculated as (Change from baseline / Baseline result *100).
rTNSS over the 14-day treatment period | Up to Day 14
  This parameter evaluates the mean change in AM rTNSS from baseline over the 14-day treatment period. The AM rTNSS is a rating of the severity of nasal symptoms over the previous 12 hours and is performed in the morning.The rTNSS was calculated as the sum of the participant-reported severity scores for nasal symptoms, and value ranged from 0 (no signs/symptoms evident) to 12 (severe signs/symptoms that is hard to tolerate).
Mean change from baseline in PM participant-reported rTNSS over the 14-day treatment period | Up to Day 14
  This parameter evaluates the mean change in PM rTNSS from baselineover the 14-day treatment period. The PM rTNSS is a rating of the severity of nasal symptoms over the previous 12 hours and is performed in the evening.The rTNSS was calculated as the sum of the participant-reported severity scores for nasal symptoms, and value ranged from 0 (no signs/symptoms evident) to 12 (severe signs/symptoms that is hard to tolerate).
Mean change from baseline in AM participant-reported iTNSS over the 14-day treatment period | Up to Day 14
  This parameter evaluates the mean change in AM iTNSS from baselineover the 14-day treatment period. The AM iTNSS is the severity rating of the instantaneous nasal symptom at a time point. The iTNSS was calculated as the sum of the participant-reported severity scores for nasal symptoms, and value ranged from 0 (no signs/symptoms evident) to 12 (severe signs/symptoms) that is hard to tolerate.
Mean change from baseline in PM participant-reported iTNSS over the 14-day treatment | Up to Day 14
  This parameter evaluates the mean change in PM iTNSS from baselineover the 14-day treatment period.The PM iTNSS is the severity rating of the instantaneous nasal symptom at a time point. The iTNSS was calculated as the sum of the participant-reported severity scores for nasal symptoms, and value ranged from 0 (no signs/symptoms evident) to 12 (severe signs/symptoms) that is hard to tolerate.
Mean change from baseline in AM participant-reported rTOSS over the 14-day treatment period | Up to Day 14
  This parameter evaluates the mean change in AM rTOSS from baselineover the 14-day treatment period.
  The AM rTOSS is a rating of the severity of ocular symptoms over the previous 12 hours and is performed in the morning.The total ocular symptom score (TOSS) is the sum of three symptom scores for itchy/burning eyes, watery eyes, and red eyes, where each symptom is scored on a scale of 0 to 3. Higher scores indicate more severe ocular symptoms, while lower scores indicate less severe ocular symptoms.
Mean change from baseline in PM participant-reported rTOSS over the 14-day treatment period | Up to Day 14
  This parameter evaluates the mean change in PM rTOSS from baselineover the 14-day treatment period.
  The PM rTOSS is a rating of the severity of ocular symptoms over the previous 12 hours and is performed in the morning.The total ocular symptom score (TOSS) is the sum of three symptom scores for itchy/burning eyes, watery eyes, and red eyes, where each symptom is scored on a scale of 0 to 3. Higher scores indicate more severe ocular symptoms, while lower scores indicate less severe ocular symptoms.
Mean change from baseline in AM participant-reported iTOSS over the 14-day treatment period | Up to Day 14
  This parameter evaluates the mean change in AM iTOSS from baselineover the 14-day treatment period.
  The AM iTOSS is the severity rating of the ocular symptom at a time point.The total ocular symptom score (TOSS) is the sum of three symptom scores for itchy/burning eyes, watery eyes, and red eyes, where each symptom is scored on a scale of 0 to 3. Higher scores indicate more severe ocular symptoms, while lower scores indicate less severe ocular symptoms.
Mean change from baseline in PM participant-reported iTOSS over the 14-day treatment period | Up to Day 14
  This parameter evaluates the mean change in PM iTOSS from baselineover the 14-day treatment period.
  The PM iTOSS is the severity rating of the ocular symptom at a time point.The total ocular symptom score (TOSS) is the sum of three symptom scores for itchy/burning eyes, watery eyes, and red eyes, where each symptom is scored on a scale of 0 to 3. Higher scores indicate more severe ocular symptoms, while lower scores indicate less severe ocular symptoms.
Mean change from baseline in the daily rTNSS | Up to Day 14
  This parameter evaluates the mean change in rTNSS (ie Day 1 measurement = Average of the PM assessment on Day 1 and AM assessment of Day 2 and so on) from baseline for each day.The rTNSS was calculated as the sum of the participant-reported severity scores for nasal symptoms, and value ranged from 0 (no signs/symptoms evident) to 12 (severe signs/symptoms that is hard to tolerate).
Mean change from baseline in the daily iTNSS | Up to Day 14
  This parameter evaluates the mean change in iTNSS (ie Day 1 measurement = Average of the PM assessment on Day 1 and AM assessment of Day 2 and so on) from baseline for each day.The iTNSS was calculated as the sum of the participant-reported severity scores for nasal symptoms, and value ranged from 0 (no signs/symptoms evident) to 12 (severe signs/symptoms that is hard to tolerate).
Mean change from baseline in the daily rTOSS | Up to Day 14
  This parameter evaluates the mean change in rTOSS (ie Day 1 measurement = Average of the PM assessment on Day 1 and AM assessment of Day 2 and so on) from baseline for each day. The total ocular symptom score (TOSS) is the sum of three symptom scores for itchy/burning eyes, watery eyes, and red eyes, where each symptom is scored on a scale of 0 to 3. Higher scores indicate more severe ocular symptoms, while lower scores indicate less severe ocular symptoms.
Mean change from baseline in the daily iTOSS | Up to Day 14
  This parameter evaluates the mean change in iTOSS (ie Day 1 measurement = Average of the PM assessment on Day 1 and AM assessment of Day 2 and so on) from baseline for each day. The total ocular symptom score (TOSS) is the sum of three symptom scores for itchy/burning eyes, watery eyes, and red eyes, where each symptom is scored on a scale of 0 to 3. Higher scores indicate more severe ocular symptoms, while lower scores indicate less severe ocular symptoms.
Mean change from baseline in the daily AM rTNSS | Up to Day 14
  This parameter evaluates the mean change in AM rTNSS from baseline for each day.The rTNSS was calculated as the sum of the participant-reported severity scores for nasal symptoms, and value ranged from 0 (no signs/symptoms evident) to 12 (severe signs/symptoms that is hard to tolerate).
Mean change from baseline in the daily PM rTNSS | Up to Day 14
  This parameter evaluates the mean change in PM rTNSS from baseline for each day.The rTNSS was calculated as the sum of the participant-reported severity scores for nasal symptoms, and value ranged from 0 (no signs/symptoms evident) to 12 (severe signs/symptoms that is hard to tolerate).
Mean change from baseline in the daily AM iTNSS | Up to Day 14
  This parameter evaluates the mean change in AM iTNSS from baseline for each day.The iTNSS was calculated as the sum of the participant-reported severity scores for nasal symptoms, and value ranged from 0 (no signs/symptoms evident) to 12 (severe signs/symptoms that is hard to tolerate).
Mean change from baseline in the daily PM iTNSS | Up to Day 14
  This parameter evaluates the mean change in PM iTNSS from baseline for each day.The iTNSS was calculated as the sum of the participant-reported severity scores for nasal symptoms, and value ranged from 0 (no signs/symptoms evident) to 12 (severe signs/symptoms that is hard to tolerate).
Mean change from baseline in the daily AM rTOSS | Up to Day 14
  This parameter evaluates the mean change in AM rTOSS from baseline for each day. The total ocular symptom score (TOSS) is the sum of three symptom scores for itchy/burning eyes, watery eyes, and red eyes, where each symptom is scored on a scale of 0 to 3. Higher scores indicate more severe ocular symptoms, while lower scores indicate less severe ocular symptoms.
Mean change from baseline in the daily PM rTOSS | Up to Day 14
  This parameter evaluates the mean change in PM rTOSS from baseline for each day. The total ocular symptom score (TOSS) is the sum of three symptom scores for itchy/burning eyes, watery eyes, and red eyes, where each symptom is scored on a scale of 0 to 3. Higher scores indicate more severe ocular symptoms, while lower scores indicate less severe ocular symptoms.
Mean change from baseline in the daily AM iTOSS | Up to Day 14
  This parameter evaluates the mean change in AM iTOSS from baseline for each day. The total ocular symptom score (TOSS) is the sum of three symptom scores for itchy/burning eyes, watery eyes, and red eyes, where each symptom is scored on a scale of 0 to 3. Higher scores indicate more severe ocular symptoms, while lower scores indicate less severe ocular symptoms.
Mean change from baseline in the daily PM iTOSS | Up to Day 14
  This parameter evaluates the mean change in PM iTOSS from baseline for each day. The total ocular symptom score (TOSS) is the sum of three symptom scores for itchy/burning eyes, watery eyes, and red eyes, where each symptom is scored on a scale of 0 to 3. Higher scores indicate more severe ocular symptoms, while lower scores indicate less severe ocular symptoms.
Mean change from baseline in individual nasal symptoms (runny nose, nasal congestion, nasal itching and sneezing) of r TNSS over the 14-day treatment period | Up to Day 14
  This parameter evaluates the mean change in individual nasal symptoms (runny nose, nasal congestion, nasal itching and sneezing) of rTNSS from baseline over the 14-day treatment period.
  The individual nasal symptoms (rhinorrhea, nasal congestion, nasal itching, and sneezing) is scored on a scale of 0 to 3, higher scores indicate more severe symptoms, while lower scores indicate less severe symptoms.
Mean change from baseline in individual nasal symptoms (runny nose, nasal congestion, nasal itching and sneezing) of AM rTNSS over the 14-day treatment period. | Up to Day 14
  This parameter evaluates the mean change in individual nasal symptoms (runny nose, nasal congestion, nasal itching and sneezing) of AM rTNSS from baseline over the 14-day treatment period.
  The individual nasal symptoms (rhinorrhea, nasal congestion, nasal itching, and sneezing) is scored on a scale of 0 to 3, higher scores indicate more severe symptoms, while lower scores indicate less severe symptoms.
Mean change from baseline in individual nasal symptoms (runny nose, nasal congestion, nasal itching and sneezing) of PM rTNSS over the 14-day treatment period. | Up to Day 14
  This parameter evaluates the mean change in individual nasal symptoms (runny nose, nasal congestion, nasal itching and sneezing) of PM rTNSS from baseline over the 14-day treatment period.
  The individual nasal symptoms (rhinorrhea, nasal congestion, nasal itching, and sneezing) is scored on a scale of 0 to 3, higher scores indicate more severe symptoms, while lower scores indicate less severe symptoms.
Mean change from baseline in individual ocular symptoms (itching/burning eyes, tearing/watering eyes, and redness eyes) of rTOSS over the 14-day treatment period | Up to Day 14
  This parameter evaluates the mean change in individual ocular symptoms (itching/burning eyes, tearing/watering eyes, and redness eyes) of rTOSS from baseline over the 14-day treatment period.
  The individual ocular symptoms (itching/burning eyes, tearing/watering eyes, and redness eyes) of rTOSS is scored on a scale of 0 to 3, higher scores indicate more severe symptoms, while lower scores indicate less severe symptoms.
Mean change from baseline in individual ocular symptoms (itching/burning eyes, tearing/watering eyes, and redness eyes) of AM rTOSS over the 14-day treatment period | Up to Day 14
  This parameter evaluates the mean change in individual ocular symptoms (itching/burning eyes, tearing/watering eyes, and redness eyes) of AM rTOSS from baseline over the 14-day treatment period.
  The individual ocular symptoms (itching/burning eyes, tearing/watering eyes, and redness eyes) of rTOSS is scored on a scale of 0 to 3, higher scores indicate more severe symptoms, while lower scores indicate less severe symptoms.
Mean change from baseline in individual ocular symptoms (itching/burning eyes, tearing/watering eyes, and redness eyes) of PM rTOSS over the 14-day treatment period | Up to Day 14
  This parameter evaluates the mean change in individual ocular symptoms (itching/burning eyes, tearing/watering eyes, and redness eyes) of PM rTOSS from baseline over the 14-day treatment period.
  The individual ocular symptoms (itching/burning eyes, tearing/watering eyes, and redness eyes) of rTOSS is scored on a scale of 0 to 3, higher scores indicate more severe symptoms, while lower scores indicate less severe symptoms.
Proportion and frequency of participants who use the rescue medication | Up to Day 14
  The proportion of participants who use the rescue medication，and the frequency of usage during the treatment.
Mean change from baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) score of general activities on day 15 | Day1, Day 8, Day 15
  Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) has 28 questions in 7 domains (activity limitation, sleep problems, nose symptoms, eye symptoms, non-nose/eye symptoms, practical problems and emotional function). Each question on a 7-point scale (0 = not impaired at all - 6 = severely impaired). The overall RQLQ score is the mean of all 28 responses.
Safety and tolerability of PG-011 Nasal Spray | Up to Day 21
  Incidence of treatment-emergent adverse events (AEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Professor, Principal Investigator — Beijing Tongren Hospital
Locations (38):
- China (38):
  - Beijing Shijitan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Youan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Gansu Provincial people's Hospital, Lanzhou, Gansu
  - The NO. 2 Hospital of Baoding, Baoding, Hebei
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Hebei Petro China Central Hospital, Langfang, Hebei
  - Hebei Provincial Hospital of Traditional Chinese Medicine, Shijiazhuang, Hebei
  - Hebei Provincial People's Hospital, Shijiazhuang, Hebei
  - Daqing people's Hospital, Daqing, Heilongjiang
  - Harbin Medical University Affiliated Fourth Hospital, Harbin, Heilongjiang
  - Luo Yang First People's Hospital, Luoyang, Henan
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Zhengzhou Central Hospital, ,, Zhengzhou, Henan
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Tonghua Central Hospital, Tonghua, Jilin
  - The central hospital of shenyang medical college, Shengyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Baotou Central Hospital, Baotou, Neimenggu
  - Chifeng Municipal Hospital, Chifeng, Neimenggu
  - Affiliated Hospital Of Inner Mongolia Medical University, Hohhot, Neimenggu
  - First People's Hospital of Yinchuan, Yinchuan, Ningxia
  - People's Hospital of Ningxia Hui autonomous region, Yinchuan, Ningxia
  - Shandong Second Provincial People's Hospital, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Yantai YuHuangDing Hospital, Yantai, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Sinopharm Tongmei General Hospital, Datong, Shanxi
  - Linfen Central Hospital, Linfen, Shanxi
  - Linfen People's Hospital, Linfen, Shanxi
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Xianyang Hospital of Yan'an University, Xianyang, Shanxi
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi’an, Shanxi
  - Xian XD Group Hospital, Xi’an, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi

IPD SHARING:
Plan to Share IPD: No